CLINICAL TRIAL: NCT02818257
Title: An Investigation Exploring Adhesive Materials and Their Ability to Handle Moisture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CP263
Record Dates: First submitted 2016-06-21; First posted 2016-06-29 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Strip A (wet) (Experimental): Six strips of Strip A are applied on skin wetted with two different buffers (3 strips each)
  Interventions: Other: Strip A
- Strip A (dry) (Experimental): Six strips of Strip A are applied on skin that is dry (3 strips) and wetted with buffer (3 strips)
  Interventions: Other: Strip A
- Strip B (wet) (Experimental): Six strips of Strip B are applied on skin wetted with two different buffers (3 strips each)
  Interventions: Other: Strip B
- Strip B (dry) (Experimental): Six strips of Strip B are applied on skin that is dry (3 strips) and wetted with buffer (3 strips)
  Interventions: Other: Strip B
- Strip C (wet) (Experimental): Six strips of Strip C are applied on skin wetted with two different buffers (3 strips each)
  Interventions: Other: Strip C
- Strip C (dry) (Experimental): Six strips of Strip C are applied on skin that is either dry (3 strips) or wetted with buffer (3 strips)
  Interventions: Other: Strip C

INTERVENTIONS:
Other: Strip A — Adhesive strip A
  Arms: Strip A (dry); Strip A (wet)
Other: Strip B — Adhesive strip B
  Arms: Strip B (dry); Strip B (wet)
Other: Strip C — Adhesive strip C
  Arms: Strip C (dry); Strip C (wet)

SUMMARY:
The aim is to investigate the impact that water absorption properties in adhesives has on adhesion.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Be at least 18 years of age and have full legal capacity
* Have intact skin on the area used in the investigation

Exclusion Criteria:

* Currently receiving or have within the past 2 month received radio- and/or chemotherapy
* Currently receiving or have within the past month received topical steroid treatment in the abdominal skin area or systemic steroid (tablet/injection) treatment.
* Are pregnant or breastfeeding
* Having dermatological problems in the abdominal area (assessed by investigator)
* Participate in other clinical investigations or have previously participated in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Peel force used to removed adhesive | 60 min
  The three strips applied to skin that has received the same treatment (either buffer 1, buffer 2 or dry) are removed at three different time points (max 60 min) and the peel force is measured.
  Peel force (90 degree angle from skin) The tensile tester was mounted on a tripod under which the subject was lying. In this way the tensile tester measures the force (Newton), which was needed to remove the adhesive from the skin with a constant speed and with a mean angel of 90°

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No